CLINICAL TRIAL: NCT00733330
Title: Computer Assisted Navigation in Minimally Invasive Total Knee Arthroplasty: Comparing the Alignment Achieved Using the DePuy Ci Minimally Invasive (Mi) Versus the DePuy Non Navigated Conventional Total Knee Arthroplasty.
Brief Title: Minimally Invasive Total Knee Replacement - Navigated Versus Non-navigated Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A sample size recalculation indicated an increase from 154 to 1500 subjects was required so the study stopped as new target was considered unfeasible.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 03/10
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty, Knee, TKA, TKR, CAS, minimally invasive
MeSH Terms: conditions — Osteoarthritis; Apraxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional TKR arm (Other): Patients to receive treatment with either a P.F.C. Sigma or L.C.S. knee using the conventional manual surgical technique
  Interventions: Device: Either P.F.C. Sigma or L.C.S. Complete knee replacement using the conventional surgical approach and manual surgical technique
- MiTKR CAS arm (Active Comparator): Patients to receive treatment with either a P.F.C. or L.C.S. knees in chronological order into the CAS group which will use minimally invasive surgery and computer navigation
  Interventions: Device: Either P.F.C. Sigma or L.C.S. Complete knee replacement using minimally invasive surgical approach and computer navigation

INTERVENTIONS:
Device: Either P.F.C. Sigma or L.C.S. Complete knee replacement using the conventional surgical approach and manual surgical technique — Orthopaedic implants for total knee replacement implanted with a standard approach using standard instrumentation
  Arms: Conventional TKR arm
Device: Either P.F.C. Sigma or L.C.S. Complete knee replacement using minimally invasive surgical approach and computer navigation — Orthopaedic implants for total knee replacement implanted with a minimally invasive approach and computer navigation
  Arms: MiTKR CAS arm

SUMMARY:
The primary objective of this investigation is to compare the precision of long leg alignment achieved by the two types of procedure. The secondary objectives of this investigation are to:

Compare the accuracy of long leg alignment achieved by the two types of procedure.

Compare the number of optimal implantations achieved by the two types of procedure.

Compare the clinical performance of the knee replacement in subjects who have undergone one of the two types of procedure.

Compare the functional outcome achieved by subjects who have undergone one of the two types of procedure.

Compare the interface radiographic appearance 5 years post-operatively between the two types of procedure.

Compare the accuracy and precision of long leg alignment achieved by the two types of procedure 5 years post-operatively, i.e., at final follow-up and also the change in accuracy and precision between the final follow-up and baseline.

Compare the Adverse Events experienced by the subjects who have undergone the two types of procedure.

DETAILED DESCRIPTION:
Primary endpoint: to compare the precision of the long leg alignment of the Ci MiTKA vs. the non navigated conventional TKA, specifically 3 months to demonstrate the variability of the mechanical axis.

Secondary endpoints: to compare the precision of the long leg alignment of the Ci MiTKA vs. the non navigated conventional TKA specifically to demonstrate the proportion of procedures that fall within a satisfactory alignment window in either group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 80 years inclusive.
* Subjects who require a primary total knee replacement and are considered by the Investigator to be suitable for the specific knee prosthesis identified in the protocol.
* Subjects who are able to give and have given voluntary, written informed consent to participate in this clinical investigation.
* Subjects who have given consent to the transfer of his/her information to DePuy.
* Subjects who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

Exclusion Criteria:

* Subjects who have a pre-operative limb deformity of equal to or greater than 10° varus or 15° valgus as defined using the anatomical axis.
* Subjects who have a fixed flexion contracture of greater than 10º.
* Subjects who are clinically obese i.e. BMI ≥30.
* Subjects who have, in the opinion of the Investigator, an existing condition that would compromise their participation and follow-up in this study.
* Female subjects who are pregnant or lactating.
* Subjects who are known drug or alcohol abusers or have a psychological disorder that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical investigation with an investigational product in the last 3 months.
* Subjects currently involved in any personal injury litigation, medical-legal or worker's compensations claims.
* Subjects who have previously had a prosthetic knee replacement device (any type) of the affected knee.
* Subjects who present with ankylosis of the hip joint on the side to be treated or previous ipsilateral Upper Tibial Osteotomy/High Tibial Osteotomy.
* Subjects who require simultaneous bilateral total knee replacements.
* Subjects who have had a contralateral TKA performed less than six months before the proposed TKA.
* Subjects who have had a contralateral TKA and that knee was previously entered in the study.
* Subjects who, in the opinion of the surgeon, will require a contralateral TKA within 6 months of the index procedure.
* Subjects in whom the surgeon intends to implant a knee component that is not one of those listed in Table 1.
* Subjects who have inflammatory arthritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Newport Orthopaedic Institute, Newport Beach, California
  - Wake Forest University, Winston-Salem, North Carolina
  - Joint Reconstruction Center, UPMC, Pittsburgh, Pennsylvania
- Sportsmed, Adelaide, South Australia, Australia
- Ascot & Mercy Hospital, Remuera, Aukland 5, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 86 subjects were enrolled at 5 sites.
Pre-assignment Details: 2 subjects were intraoperatively excluded and did not receive surgery.
Groups:
- MiTKR CAS Arm: Either a P.F.C. or L.C.S. using minimally invasive surgery and computer navigation
- Conventional TKR Arm: Either a P.F.C. Sigma or L.C.S. knee using the conventional manual surgical technique
Period: Overall Study
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Started | 32 | 52
Completed | 30 | 48
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: 86 subjects were enrolled, but 2 were intraoperatively excluded and did not receive surgery. Gender data is unavailable on one MiTKR subject.
Groups:
- Total: Total of all reporting groups
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm | Total
Number analyzed (Participants) | 32 | 52 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (6.3) | 65.5 (8.8) | 65.8 (7.9)
Gender [Number; unit: participants]
  Female | 18 | 31 | 49
  Male | 13 | 21 | 34
Region of Enrollment [Number; unit: participants]
  United States | 16 | 26 | 42
  Australia | 9 | 12 | 21
  New Zealand | 7 | 14 | 21

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Precision of the Long Leg Alignment Between the Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: Alignment will be measured on long leg weight bearing X-rays performed when the subject has full leg extension (+/-5 degrees)
Time Frame: 6 - 12 Weeks
Population: The study was terminated before completion due to business purposes, therefore no radiographs were analyzed.
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Compare the Proportion of Procedures That Fall Within a Satisfactory Alignment Window Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: An independent radiographic observer will determine and record alignment.
Time Frame: operative
Population: The study was terminated before completion due to business purposes, therefore no radiographs were analyzed and there are no results for this outcome.
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Compare the Number of Optimal Implantations Achieved From Pre-op to 6-12 Weeks Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: Achieved alignment results will be measured on post-op X-rays taken at the time the subject has achieved full extension.
Time Frame: 4 - 12 Weeks
Population: as for outcome 2
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
Time Frame: Pre-op
Population: Of the 84 subjects who received surgery, there were 3 missing outcomes for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 31 | 50
points | 54.1 (16) | 45.3 (13.8)

5. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: The American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
Time Frame: 4 Weeks
Population: There were 19 missing outcomes and 1 consent withdrawal for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 20 | 44
points | 63.8 (19.5) | 66.3 (16.6)

6. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 4
Time Frame: 8 Weeks
Population: There were 19 missing outcomes, 1 consent withdrawal, 1 Lost to Follow Up and 1 protocol violation for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 20 | 42
points | 78.8 (16.8) | 77.5 (15.6)

7. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 4
Time Frame: 12 Weeks
Population: There were 32 missing outcomes, 1 consent withdrawal, 2 Lost to Follow Up and 1 protocol violation for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 13 | 35
points | 85.5 (17.5) | 80.9 (15.1)

8. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 4
Time Frame: 6 Months
Population: There were 10 missing outcomes, 1 consent withdrawal, 2 Lost to Follow Up and 1 protocol violation for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 22 | 48
points | 83.3 (18.2) | 84.6 (15.1)

9. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 4
Time Frame: 1 year
Population: There were 22 missing outcomes, 1 consent withdrawal, 2 Lost to Follow Up, and 3 protocol violations for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 17 | 39
points | 86.5 (13.4) | 89.6 (11.5)

10. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 4
Time Frame: 2 years
Population: There were 41 missing outcomes, 1 consent withdrawal, 2 Lost to Follow Up, and 3 protocol violations for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 7 | 30
points | 76.4 (20.5) | 87.5 (10.2)

11. Secondary Outcome: To Compare American Knee Society Knee Score Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 4
Time Frame: 5 years
Population: The study was terminated before completion due to business purposes, therefore no outcomes are available for this endpoint.
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: The Oxford Knee Score (OKS) is a 12 to 60 point patient reported outcome (PRO) score (where 12 indicates the best outcome) that evaluates the affected knee. The total score is composed of Pain and Function.
Time Frame: pre-op
Population: There were 2 missing outcomes for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 31 | 51
points | 33.4 (8.0) | 36.1 (7.4)

13. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 12
Time Frame: 4 Weeks
Population: There were 19 missing outcomes and 1 consent withdrawal for this outcome.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 19 | 45
points | 32.3 (10.2) | 31.4 (7.5)

14. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 12
Time Frame: 8 Weeks
Population: There were 19 missing outcomes, 1 consent withdrawal, 1 protocol violation, and 1 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 20 | 42
points | 24.7 (7.2) | 26.5 (8.5)

15. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 12
Time Frame: 12 Weeks
Population: There were 33 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 2 Lost to Follow up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 12 | 35
points | 20.2 (7.6) | 23.7 (7.0)

16. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 12
Time Frame: 6 Months
Population: There were 10 missing outcomes, 1 protocol violation, 1 consent withdrawal and 2 Lost to Follow up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 22 | 48
points | 20.0 (8.4) | 20.2 (7.0)

17. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 12
Time Frame: 1 Year
Population: There were 21 missing outcomes, 3 protocol violations, 1 consent withdrawal, and 2 Lost to Follow up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 17 | 40
points | 16.5 (5.1) | 17.5 (6.1)

18. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 12
Time Frame: 2 years
Population: There were 41 missing outcomes, 3 protocol violations, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 7 | 30
points | 17.0 (6.6) | 17.8 (7.5)

19. Secondary Outcome: To Compare Oxford Knee Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 12
Time Frame: 5 years
Population: The study was terminated before completion due to business purposes, therefore there are no results for this outcome.
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: WOMAC is a patient reported outcome (PRO) that evaluates the condition of subject's with knee osteoarthritis, and includes pain (score range 0-20), stiffness (score range 0-8), and physical function (score range 0-68) of the joint, where a lower score indicates a better outcome. The WOMAC total score is a combination of the three domains (pain, stiffness, and physical function) with a range of 0-96.
Time Frame: pre-op
Population: There were 4 missing outcomes for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 30 | 50
points | 34.7 (14.9) | 39.3 (14.0)

21. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 20
Time Frame: 4 Weeks
Population: There were 21 missing outcomes and 1 consent withdrawal for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 19 | 43
points | 26.2 (19.2) | 27.6 (16.5)

22. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 20
Time Frame: 8 weeks
Population: There were 22 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 1 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 19 | 40
points | 14.2 (11.5) | 18.5 (14.1)

23. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 20
Time Frame: 12 weeks
Population: There were 36 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 12 | 32
points | 14.5 (15.5) | 13.7 (11.9)

24. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 20
Time Frame: 6 months
Population: There were 16 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 22 | 42
points | 7.2 (10.4) | 7.0 (8.7)

25. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 20
Time Frame: 1 year
Population: There were 25 missing outcomes, 3 protocol violations, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 16 | 37
points | 5.9 (9.0) | 6.6 (8.5)

26. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 20
Time Frame: 2 years
Population: There were 44 missing outcomes, 3 Protocol Violations, 1 Consent Withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 5 | 29
points | 4.6 (5.8) | 6.6 (10.0)

27. Secondary Outcome: To Compare WOMAC Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 20
Time Frame: 5 years
Population: The study was terminated early for business reasons therefore there are no outcomes for this endpoint.
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: To Compare VAS Pain Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: A 100-mm visual analog scale (VAS) was used to assess pain after the subject completes the 6-minute walk test. It asks the subject to place a vertical mark on a 100-mm horizontal line, with 'No pain' listed on the left (at 0 mm) and 'Very severe pain' labeled on the right (at 100 mm). The subject is instructed to indicate the amount of pain they feel in their knee joint.
Time Frame: pre-op
Population: There were 3 missing outcomes for this endpoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 31 | 50
millimeters | 17.4 (19.8) | 24.7 (24.9)

29. Secondary Outcome: To Compare VAS Pain Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 28
Time Frame: 4 Weeks
Population: There were 23 missing outcomes and 1 Consent Withdrawal for this endpoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 18 | 42
millimeters | 10.3 (17.8) | 15.8 (23.4)

30. Secondary Outcome: To Compare VAS Pain Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 28
Time Frame: 8 Weeks
Population: There were 26 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 1 Lost to Follow up for this endpoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 20 | 35
millimeters | 8.4 (16.8) | 7.9 (13.3)

31. Secondary Outcome: To Compare VAS Pain Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 28
Time Frame: 12 Weeks
Population: There were 37 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 13 | 30
millimeters | 10.0 (17.7) | 7.5 (12.5)

32. Secondary Outcome: To Compare VAS Pain Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 28
Time Frame: 6 months
Population: There were 12 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 22 | 46
millimeters | 4.8 (11.8) | 2.9 (6.0)

33. Secondary Outcome: To Compare Interface Radiographic Appearance Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: An independent radiographer will observe and record alignment.
Time Frame: 5 years
Population: as for outcome 2
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: To Compare the Change From 6-12 Weeks & 5 Years on Long Leg Alignment.
Description: An independent radiographer will observe and record alignment
Time Frame: 5 years
Population: as for outcome 2
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: To Compare 6 Minute Walk Test Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: This score records the total distance walked (measured in feet) in 6 minutes (this time includes any time that the subject needs to stop and rest). Pre-operatively, the subject must complete both a practice walk and a test walk.
Time Frame: pre-op
Population: There were 5 missing outcomes for this endpoint.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 31 | 48
Feet | 1094.1 (326) | 990.6 (386)

36. Secondary Outcome: To Compare 6 Minute Walk Test Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: This score records the total distance walked (measured in feet) in 6 minutes (this time includes any time that the subject needs to stop and rest).
Time Frame: 4 weeks
Population: There were 21 missing outcomes and 1 consent withdrawal for this endpoint.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 18 | 44
Feet | 948.4 (395) | 922.5 (391)

37. Secondary Outcome: To Compare 6 Minute Walk Test Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 36
Time Frame: 8 weeks
Population: There were 20 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 1 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 20 | 41
Feet | 1249.9 (402) | 1079.4 (382)

38. Secondary Outcome: To Compare 6 Minute Walk Test Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 36
Time Frame: 12 weeks
Population: There were 32 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 13 | 35
Feet | 1287.1 (410) | 1259.5 (588)

39. Secondary Outcome: To Compare 6 Minute Walk Test Scores Between Subjects Who Have Undergone Minimally Invasive vs. Conventional Total Knee Arthroplasty.
Description: as for outcome 36
Time Frame: 6 months
Population: There were 13 missing outcomes, 1 protocol violation, 1 consent withdrawal, and 2 Lost to Follow Up for this endpoint.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Number analyzed (Participants) | 22 | 45
Feet | 1403.9 (442) | 1393.7 (470)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline through December 2008.
Arm/Group | MiTKR CAS Arm | Conventional TKR Arm
Serious Adverse Events (participants affected / at risk) | 2/32 | 9/52
Other Adverse Events (participants affected / at risk) | 4/32 | 7/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiTKR CAS Arm (N=32) | Conventional TKR Arm (N=52)
Nervous System Disorder (Nervous system disorders) | 0 (0) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiTKR CAS Arm (N=32) | Conventional TKR Arm (N=52)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Pain (General disorders) | 0 (0) | 3 (3)
Joint Injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
DePuy reserves the right to review the contents of publications in advance.The PI may freely disclose the trial results only after DePuy has been given the opportunity of reviewing the proposed results communications at least 30 days prior to the intended release.DePuy will advise the PI of any perceived errors,omissions or corrections but the PI will retain final editorial control.In case of disagreement,DePuy and the PI will make every effort to meet in order to discuss and resolve any issues.